CLINICAL TRIAL: NCT06355050
Title: Ultrahypofractionated, Adaptive Radiation Therapy of Prostate Cancer - Ultra-HART
Brief Title: Ultrahypofractionated, Adaptive Radiation Therapy of Prostate Cancer
Acronym: ultraHART
Status: Not yet recruiting | Type: Observational
Sponsor: Jena University Hospital (Other)
Collaborators: University Hospital Schleswig-Holstein (Other); Klinikum Stuttgart (Other); University Medical Center Göttingen (Unknown); Kantonsspital Aarau (Other); Hirslanden Stephanshorn (Unknown); Universitätsklinik Würzburg (Unknown); Radiologische Allianz Hamburg (Unknown)
Responsible Party: Principal Investigator, Georg Wurschi, Principal Investigator, Jena University Hospital
Other Study IDs: UKJ-ultraHART
Record Dates: First submitted 2024-03-27; First posted 2024-04-09 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Prostate Cancer; Adaptive Radiotherapy; Quality of Life
Keywords: Adaptive Radiotherapy; Quality of Life; Ultra-hypofractionation
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients receiving ultrahypofractionated radiotherapy
- Retrospective reference cohort: reference cohort of patients who underwent normofractionated radiotherapy or moderately hypofractionated radiotherapy earlier.
  matching 1:1:1 by tumor stage and risk profile (d'Amico)

SUMMARY:
In this prospective, multi-center cohort study, the tolerability and quality of life during ultrahypofractionated radiotherapy (RT) of early stage prostate cancer is surveyed at several institutions in Germany. Radiotherapy is delivered by an online-adaptive RT device (Varian Ethos), which is able to correct daily variations in anatomy and to adjust the irradiation plan accordingly. A digital patient questionnaire is used to asses quality of life longitudinally. Quality of life (QoL) and toxicity profiles will be correlated with planning parameters and compared to retrospective cohorts of patients who underwent normofractionated RT or moderately hypofractionated RT, respectively.

ELIGIBILITY:
Inclusion Criteria:

* no androgen deprivation therapy within the last 2 months prior to RT
* good performance status (Eastern Cooperative Oncology Group, ECOG, 0/1)
* no secondary malignancy

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * low / intermediate risk prostate cancer
  * prostate volume < 100 ccm
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2032-09-30 (Estimated)

PRIMARY OUTCOMES:
Quality of Life (EPIC 26) | longitudinally: before + during RT and during follow up (5 years, at least bi-annually)
  Expanded Prostate Cancer Index Composite 26 (questionnaire)

SECONDARY OUTCOMES:
Toxicity (CTCAE v5.0) | longitudinally: before + during RT and during follow up (5 years, at least bi-annually)
  Common Terminology Criteria for Adverse Events v5.0
Planning parameters | for every fraction, total: 5x (1 week)
  Dose constraints per organ, Conformity Indices, Quality of adaptive planning
Dose constraints | for every fraction, total: 5x (1 week)
  Dose constraints for organs at risk and target volumes per fraction
Conformity indices | for every fraction, total: 5x (1 week)
  Conformity indices for target volumes, per fraction
Quality of adaptive planning | for every fraction, total: 5x (1 week)
  Semi-quantitative score to evaluate the quality of the adaptive plan and if revisions would be required
PSA-value | longitudinally: before + during RT and during follow up (5 years, at least bi-annually)
  endpoint: Prostate-specific antigene (PSA)-recurrence free survival
Overall survival | 5 Years
Recurrence free survival | 5 Years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiotherapy and Radiation Oncology, Jena University Hospital, Jena, Germany

IPD SHARING:
Plan to Share IPD: No